CLINICAL TRIAL: NCT05931770
Title: The Effect of Child Choice With Accompanying Parent on Pediatric Anxiety and Postoperative Delirium During Induction of Anesthesia During Day Case Surgeries.
Brief Title: The Effect of Child Choice With Accompanying Parent on Postoperative Delirium During Induction of Anesthesia
Status: Completed | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 06-2023/11
Record Dates: First submitted 2023-06-25; First posted 2023-07-05 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-06

CONDITIONS: Anxiety State; Child Behavior; Postoperative Delirium
Keywords: day- case surgery, anxiety children; Postoperative Delirium
MeSH Terms: conditions — Anxiety Disorders; Child Behavior; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Child Preference: The children will prefer parents (mother or father) who will accompany them in the preoperative holding area and at induction
  Interventions: Procedure: Selection of parent(mother or father) according to children preference
- Group Parent's Preference: Parents will decide among themselves and prefer the parents (mother or father) who will accompany them from the side of the parent, in the pre-operative waiting area and during induction.
  Interventions: Procedure: Parent (mother or father) selection according to parents' preference

INTERVENTIONS:
Procedure: Selection of parent(mother or father) according to children preference — The parent who will accompany the child during the perioperative period will be determined by the child. will be determined by children preference
  Groups: Group Child Preference
Procedure: Parent (mother or father) selection according to parents' preference — Accompanying parentwho will accompany during the perioperative period will be determined by the parents. to be determined by
  Groups: Group Parent's Preference

SUMMARY:
Induction of anesthesia can be distressing both for children and their parents. Nonpharmacological behavioral interventions can reduce the anxiety of children without significant adverse effects as seen with sedative drugs.

The aim of this study will be to evaluate whether the children's or parental preference with attending parent affects on the postoperative delirium of the children or not. The delirium of the children will be assessed by the Pediatric Anesthesia Occurrence Delirium Scale (PAED)

DETAILED DESCRIPTION:
Anesthetic induction can be one of the most stressful experiences for the child during the perioperative period, with almost 50% of the children showing significant anxiety. . To minimize the effect of anxiety, several methods have been adopted, such as the introduction of day-case surgery, parental presence at the induction of anesthesia, distractions and the use of pharmacological agents like midazolam to reduce anxiety. Although the effect of parental presence on the anxiety of children and parents was studied in various studies. Whether the children's choice of parental selection affects anxiety and postoperative delirium not studied yet. In this study, we will evaluate the anxiety of children by using mYPAS and postoperative delirium by using PAED.

ELIGIBILITY:
Inclusion Criteria:

1. 5-12 years aged children
2. ASA physical Status I-II
3. Who underwent day-case surgeries in the Ear Nose and Throat Clinic

Exclusion Criteria:

1. Mentally challenged
2. Deaf Child
3. Cerebral Palsy
4. Premedicated Child
5. Language Problem
6. Unco-operative
7. Previous surgery or anesthesia history

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study included 80 children of both genders, aged 5-12 years, who underwent day-case surgeries in the Ear Nose and Throat Clinic with ASA physical Status I-II will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Evaluation with Pediatric Anesthesia Emergence Delirium Scale (PAED) in the postoperative waiting room | Postoperative 1st day
  Incidence of post-anesthesia and postoperative delirium Discordant behaviors assessed with Pediatric Anesthesia Emergence Delirium Scale (PAED) with five features, each scored using a 5-point Likert scale

SECONDARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale (mYPAS) of the children undergoing elective surgery under general anesthesia. | Perioperative period
  The mYPAS will be used to evaluate the anxiety level of children. The mYPAS is an observational measure of preoperative anxiety consisting of 27 items in 5 domains (activity, emotional expressivity, state of arousal, vocalization, and use of parents). The adjusted mYPAS total score ranges from 22.9 to 100, with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Yücedağ, Assist Prof, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)